CLINICAL TRIAL: NCT07347522
Title: Associations Between Body Composition, Energy Availability, and Lifestyle Factors in Reserve Officer Training Corps Cadets
Brief Title: Body Composition and Lifestyle Factors in ROTC
Status: Recruiting | Type: Observational
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Michael J. Ormsbee, Director of the Institute of Sports Sciences and Medicine, Florida State University
Other Study IDs: STUDY00006460
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Low Energy Availability; Physical Performance; Nutrition
Keywords: body composition; energy availability; physical fitness; Reserve Officer Training Corp; nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Reserve Officer Training Corps Cadets: Low Energy Availability or Non-Low Energy Availability

SUMMARY:
This study aims to investigates the relationships between body composition, sleep, diet, and physical fitness in ROTC cadets. Further, it aims to evaluate the accuracy of body composition screening methods and identify lifestyle factors linked to performance. Methods include body composition testing, surveys, accelerometry, and fitness score collection from cadets.

DETAILED DESCRIPTION:
This study focuses on understanding health and performance among students enrolled in Reserve Officers' Training Corps (ROTC). ROTC cadets are a population expected to maintain both academic and military-readiness demands. Many cadets must balance early-morning training, full course loads, part-time jobs, and social obligations, all of which can influence their sleep habits, nutrition choices, and physical fitness. At the same time, the assessment of body composition is an important part of military standards, yet the tools used to evaluate it vary widely and may not always reflect an individual's true physiological status. To explore these interconnected factors, this study examines patterns in cadets' body composition alongside their dietary practices, sleep behaviors, and physical fitness. By doing so, it seeks to clarify how everyday lifestyle factors may support or hinder readiness and whether commonly used body composition screening methods align with more precise measurements. Ultimately, the goal is to provide a clearer picture of the health challenges and needs of ROTC cadets and to help inform strategies that promote performance, well-being, and long-term resilience in this unique group.

ELIGIBILITY:
Inclusion Criteria:

* currently enrolled as a Reserve Officer Training Corps Cadets
* 18 years or older

Exclusion Criteria:

* pregnancy
* injuries preventing full participation in ROTC training or activities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Current members of local Reserve Officer Training Corps Cadets (ROTC) programs.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Energy Availability | 7 days
Physical Fitness | Day of study enrollment

SECONDARY OUTCOMES:
Subjective Sleep | Day of study enrollment
Body Composition | Day of study enrollment
Muscle quality | day of study enrollment
  Ultrasound echo intensity and muscle thickness
Nutrition Knowledge | day of study enrollment
  Knowledge of nutrition based on survey scores

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Sports Sciences and Medicine, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided